CLINICAL TRIAL: NCT05170282
Title: Deep Learning Magnetic Resonance Imaging Radiomics for Diagnostic Value of Hepatic Tumors in Infants
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: West China Hospital (Other)
Responsible Party: Principal Investigator, Yuhan Yang, Doctor of Medicine, West China Hospital
Other Study IDs: HX2021-345
Record Dates: First submitted 2021-12-08; First posted 2021-12-27 (Actual); Last update posted 2021-12-27 (Actual); Status verified 2021-12

CONDITIONS: Hepatoblastoma; Hepatic Hemangioendothelioma
MeSH Terms: conditions — Hepatoblastoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Retrospective cohort: The internal cohort was retrospectively enrolled in West China Hospital, Sichuan University from June 2010 and December 2020. It is a training and internal validation cohort.
  Interventions: Diagnostic Test: Radiomic Algorithm
- Prospective cohort: The same inclusion/exclusion criteria were applied for the same center prospectively. It is an external validation cohort.
  Interventions: Diagnostic Test: Radiomic Algorithm

INTERVENTIONS:
Diagnostic Test: Radiomic Algorithm — Different radiomic, machine learning, and deep learning strategies for radiomic features extraction, sorting features and model constriction.

SUMMARY:
Hepatic tumors in the perinatal period are associated with significant morbidity and mortality in affected patients. The conventional diagnostic tool, such as alpha-fetoprotein (AFP) shows limited value in diagnosis of infantile hepatic tumors. This retrospective-prospective study is aimed to evaluate the diagnostic efficiency of the deep learning system through analysis of magnetic resonance imaging (MRI) images before initial treatment.

DETAILED DESCRIPTION:
Hepatic tumors seldom occur in the perinatal period. They comprise approximately 5% of the total neoplasms of various types occurring in the fetus and neonate. Infantile hemangioendothelioma is the leading primary hepatic tumor followed by hepatoblastoma. It should be mentioned that alpha-fetoprotein (AFP) is highly elevated during the first several months after birth even in normal infants, thus the diagnostic value of AFP is limited for infantile patients with hepatic tumors. This study is a retrospective-prospective design by West China Hospital, Sichuan University, including clinical data and radiological images. A retrospective database was enrolled for patients with definite histological diagnosis and available magnetic resonance imaging (MRI) images from June 2010 and December 2020. The investigators have constructed a deep learning radiomics diagnostic model on this retrospective cohort and validated it internally. A prospective cohort would recruit infantile patients diagnosed as liver tumor since January 2021. The proposed deep learning model would also be validated in this prospective cohort externally. The established model would be able to assist diagnosis for hepatic tumor in infants.

ELIGIBILITY:
Inclusion Criteria:

* Age between newborn and 12 months
* Receiving no treatment before diagnosis
* With written informed consent

Exclusion Criteria:

* Clinical data missing
* Unavailable MRI images
* Without written informed consent

Ages: 0 Months to 12 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Patients who had liver tumor and completed the abdominal MRI examination before operation, biopsy, neoadjuvant chemotherapy, and radiotherapy.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2021-01-01 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
The diagnostic accuracy of infantile liver tumors with deep learning algorithm | 1 month
  The diagnostic accuracy of infantile liver tumors with deep learning algorithm.

SECONDARY OUTCOMES:
The diagnostic sensitivity of infantile liver tumors with deep learning algorithm | 1 month
  The diagnostic sensitivity of infantile liver tumors with deep learning algorithm.
The diagnostic specificity of infantile liver tumors with deep learning algorithm | 1 month
  The diagnostic specificity of infantile liver tumors with deep learning algorithm.
The diagnostic positive predictive value of infantile liver tumors with deep learning algorithm | 1 month
  The diagnostic positive predictive value of infantile liver tumors with deep learning algorithm.
The diagnostic negative predictive value of infantile liver tumors with deep learning algorithm | 1 month
  The diagnostic negative predictive value of infantile liver tumors with deep learning algorithm.

CONTACTS AND LOCATIONS:
Locations (1):
- West China Hospital, Sichuan University, Chengdu, Sichuan, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Yang Y, Zhou Z, Li Y. MRI-based deep learning model for differentiation of hepatic hemangioma and hepatoblastoma in early infancy. Eur J Pediatr. 2023 Oct;182(10):4365-4368. doi: 10.1007/s00431-023-05113-x. Epub 2023 Jul 18. PMID 37462798